CLINICAL TRIAL: NCT05529420
Title: Interindividual Variability in Duration of Action of Rocuronium in Pediatric Patients: a Prospective Observational Study
Brief Title: Interindividual Variability in Duration of Action of Rocuronium in Pediatric Patients
Acronym: DurAct
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, Clinical Professor, Brno University Hospital
Other Study IDs: KDAR FN Brno DurAct
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2022-09

CONDITIONS: Muscle Relaxation
Keywords: duration; muscle relaxant; rocuronium
MeSH Terms: conditions — Muscle Hypotonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric patients rocuronium: In pediatric patients undergoing a planned general anesthesia with non-depolarizing muscle relaxants, induction of anesthesia will involve either standard intravenous (an opioid, anesthetic, muscle relaxant) or inhalational agents according to the preference of the anesthesiologist.
  Interventions: Other: measurement of the depth of neuromuscular blockade

INTERVENTIONS:
Other: measurement of the depth of neuromuscular blockade — time of TOF 1 measurement (= clinical effect, stimulation of the ulnar nerve - adductor pollicis muscle tension) will be documented in the CRF and if there is no need to add further doses of the muscle relaxant, TOF 2, TOF 3, TOF 4, and TOF-R ≥ 0,9 (= time to full recovery from the effect of the non-depolarizing muscle relaxant) will also be registered.
  Other Names: neuromuscular blockade depth

SUMMARY:
Muscle relaxants represent an important part of general anesthesia in adult and pediatric patients. Their role is to facilitate intubation and enable some surgical interventions.

At our workplace, monitoring of the depth of neuromuscular blockade is a standard procedure in accordance with the 2017 recommendation of ČSARIM entitled "Principles of Patient Safety in Anesthesiology" [1,2]. At present, we mainly use rocuronium. One of the advantages of this non-depolarizing steroidal muscle relaxant with a rapid onset and intermediate duration of action is the existence of the specific antagonist sugammadex.

DETAILED DESCRIPTION:
Given the observational study design, we expect that no informed consent will be required. In pediatric patients undergoing a planned general anesthesia with non-depolarizing muscle relaxants, induction of anesthesia will involve either standard intravenous (an opioid, anesthetic, muscle relaxant) or inhalational agents according to the preference of the anesthesiologist. Standard monitoring during general anesthesia will be carried out including measurement of the depth of neuromuscular blockade (Train of Four, TOF, Avance CS2 machine, relaxometry module, stimulating current of 50 mA) every minute and body temperature monitoring. Subsequently, these parameters including the age-related minimum alveolar concentration of sevoflurane will be documented in the Case Report Form (CRF).

Rocuronium will be administered at a dose according to the Summary of Product Characteristics (SPC) and local expertise. Patient demographic parameters, dose of rocuronium, time of its administration, and time of TOF 1 measurement (= clinical effect, stimulation of the ulnar nerve - adductor pollicis muscle tension) will be documented in the CRF and if there is no need to add further doses of the muscle relaxant, TOF 2, TOF 3, TOF 4, and TOF-R ≥ 0,9 (= time to full recovery from the effect of the non-depolarizing muscle relaxant) will also be registered. In addition, reversal of neuromuscular blockade if applicable and the Aldrete score in the first and fifth minute after extubation will be recorded.

In patients monitored after an intervention in a recovery room, possible complications occurring within at least 30 minutes postoperatively will be documented (desaturation, the need for oxygen therapy, tachycardia >150 beats per minute, bradycardia <50 beats per minute, aspiration, sore throat, cough, hoarseness). All patients will be screened for aspiration pneumonia on chest X-ray within the first 24 hours after an intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 0 to 18 years admitted for a planned intervention in general anesthesia with orotracheal or nasotracheal intubation and use of the muscle relaxant rocuronium
* ASA score 1 or 2

Exclusion Criteria:

* Patients requiring more types of muscle relaxants during general anesthesia induction
* Patients requiring a rapid sequence induction to general anesthesia
* Neuromuscular disease
* Concomitant medication interfering with the metabolism of muscle relaxants (anticonvulsants, aminoglycosides, polypeptide antibiotics)
* Comorbidities - renal or hepatic disorders
* ASA ≥ 3

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients aged 0 to 18 years admitted for a planned intervention in general anesthesia with orotracheal or nasotracheal intubation and use of the muscle relaxant rocuronium
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Age-based TOF 1 recovery | intraoperatively
  Comparison of duration of clinical action after single-dose rocuronium to TOF 1 in different pediatric age groups

SECONDARY OUTCOMES:
TOF 1 recovery | Intraoperatively
  Comparison of duration of clinical action after single-dose rocuronium to TOF 1 relative to patient weight, gender, and height
Muscle relaxation recovery time characteristics | Intraoperatively
  Comparison of interval from single-dose rocuronium to TOF 2, 3, and 4 in different pediatric age groups and relative to patient weight, gender, and height
Time to full muscle relaxation recovery | Intraoperatively
  Comparison of interval from single-dose rocuronium to full recovery in different pediatric age groups and relative to patient weight, gender, and height
Muscle relaxation reversal | Intraoperatively
  Identification of a patient subgroup requiring antagonization after a surgical procedure
Postoperative complications | 24 hours postoperatively
  Monitoring of postoperative complications of general anesthesia
Impact of sevoflurane anesthesia on the pharmacodynamics of rocuronium | intraoperatively
  Influence of sevoflurane concentration on rocuronium pharmacodynamics
Impact of body temperature on pharmacodynamics of rocuronium | intraoperatively
  Influence of temperature on rocuronium pharmacodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Petr Stourac, prof. MD., Ph.D., MBA, Study Chair — Department of paediatric anaesthesia and intensive care medicine
Locations (1):
- Brno University Hospital, Brno, South Moravian, Czechia

IPD SHARING:
Plan to Share IPD: Undecided